CLINICAL TRIAL: NCT01991106
Title: A Multi-centre Randomized Controlled Trial Examining the Effects of High Intensity Interval Training on Cardio-metabolic Outcomes in Obese Children and Adolescents
Brief Title: Effects of Exercise Intensity in Obese Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009/1313
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: Exercise; Myocardial function; Vascular function; Cardiovascular disease/prevention & control; Paediatric obesity; Visceral adipose tissue
MeSH Terms: conditions — Obesity; Motor Activity; Cardiovascular Diseases | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High intensity interval training (Experimental): 10-minute warm up at 60-70% of maximal heart rate (HRmax). Then walking, running or cycling at 85-95% of maximal heart rate at intervals of 4 x 4 minutes, with 3 minute active breaks (50-70% of HRmax) between intervals. A 5-minute cool down period.
  Interventions: Behavioral: High intensity interval training; Dietary Supplement: Nutritional advice
- Moderate intensity continuous training (Experimental): walking, running or cycling continuously at 60-70% HRmax for 44 minutes.
  Interventions: Behavioral: Moderate intensity continuous training; Dietary Supplement: Nutritional advice
- nutritional advice (Active Comparator): 10 individual nutrition consultations with an accredited dietitian over the 12 month period. Content of consultations will include healthy food choices, portion sizes and regular mealtimes.
  Interventions: Dietary Supplement: Nutritional advice
- non-obese children (No Intervention): 100 healthy non-obese children aged 7-16 (controls)

INTERVENTIONS:
Behavioral: High intensity interval training — Twelve weeks of 2-3 supervised training sessions each week.
  Other Names: HIIT
  Arms: High intensity interval training
Behavioral: Moderate intensity continuous training — Twelve weeks of 2-3 supervised training sessions each week.
  Other Names: MICT
  Arms: Moderate intensity continuous training
Dietary Supplement: Nutritional advice — healthy food choices, portion sizes and regular mealtimes
  Arms: High intensity interval training; Moderate intensity continuous training; nutritional advice

SUMMARY:
The prevalence of paediatric obesity has increased over the last two decades and with it, an increased diagnosis of lifestyle-related diseases in children and adolescents. High intensity interval training has recently been explored as an alternate to traditional aerobic exercise in adults with chronic disease and has potential to induce rapid reversal of subclinical disease markers in obese children and adolescents.

High intensity interval training has recently been explored as an alternate to traditional aerobic exercise in adults with chronic disease and has potential to induce rapid reversal of subclinical disease markers in obese children and adolescents.

Goal: The primary aim of this randomised controlled trial is to evaluate the effectiveness of a high intensity interval training intervention on myocardial function, vascular function and visceral adipose tissue in obese children and adolescents at baseline, three and twelve months.

Method: Multi-centre randomised controlled trial of 100 obese children and adolescents in the cities of Trondheim (Norway) and Brisbane (Australia). Participants will be randomised to (1) high intensity interval training, (2) moderate intensity continuous training or (3) nutrition advise. Participants will partake in supervised exercise training and/or nutrition consultations for 3 months. Measurements for all study endpoints will occur at baseline, 3 months (post intervention) and 12 months (follow up).

Scientific Significance : This randomised controlled trial will general substantial information regarding the effects of exercise intensity on paediatric obesity, specifically the cardio-metabolic health of this at-risk population. It is expected that communication of results will allow for more robust and realistic guidelines regarding exercise prescription in this population to be formed while outlining the benefits of high intensity interval training on subclinical markers of disease.

DETAILED DESCRIPTION:
Worldwide, childhood overweight and obesity rates are approximately 10%, this high incidence attributed to a physically inactive lifestyle and inappropriate nutrition. Early cohort studies illustrated that fifty per cent of obese children became obese adults and consequently had an higher risk for metabolic syndrome than obese adults who were not obese as children. Both female and male overweight children and adolescents had a 30% increase in all cause mortality. The increases in risk of death were independent of adult body mass index.

Systematic reviews suggest that lifestyle and exercise interventions in obese children and adolescents can lead to improvements in anthropometric and cardio-metabolic outcomes, but these are not inclusive of several important outcomes such as myocardial and vascular function or visceral adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

- Obese (BMI ≥ 95th percentile - age and sex specific criteria)

Exclusion Criteria:

* Elevated blood pressure (≥ 95th percentile for systolic or diastolic values)
* Congenital heart disease
* Coronary artery disease
* Family history of hypertropic obstructive cardiomyopathy
* Any abnormality during rest or stress echocardiography which indicates it would be unsafe to participate
* Self reported kidney failure
* Any major organ transplant
* Considerable pulmonary disease including severe or poorly controlled asthma
* Smoking
* Diabetes
* Epilepsy or a history of seizures
* Orthopaedic or neurological limitations to exercise
* Diagnosed attention deficit hypersensitivity disorder
* Steroid medications
* Participation in another research study

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Peak systolic tissue velocity | 12 weeks
  systolic tissue Doppler velocity assessed during resting and stress echocardiography

SECONDARY OUTCOMES:
Subcutaneous and total abdominal adipose tissue | 12 weeks, 12 months
  Assessed using MRI
Cardiorespiratory fitness (VO2peak) | 12 weeks, 12 months
  Assessed using a maximal treadmill test
Body composition | 12 weeks, 12 months
  Assessed using DXA (UQ), BodPod (NTNU)
Blood biochemistry | 12 weeks, 12 months
  Analysed for lipids, glucose, insulin, inflammatory makers, satiety hormones, oxidative stress
Physical activity | 12 weeks, 12 months
  Assessed through 7 day accelerometry
Dietary analysis | 12 weeks, 12 months
  Assessed through a three-day food record
Myocardial structure and cardiac adipose tissue (UQ) | 12 weeks
  Assessed through cardiac MRI; participants > 12 years only
Arterial stiffness | 12 weeks, 12 months
  Assessed through pulse wave velocity and pulse wave analysis
Autonomic function | 12 weeks, 12 months
  Assessed through heart rate variability and heart rate recovery
Quality of life | 12 weeks, 12 months
  Assessed through the Paediatric Quality of Life Inventory
Visceral adipose tissue | 12 weeks, 12 months
  assessed by magnetic resonance imaging (MRI)
Vascular function | 12 weeks, 12 months
  Assessed through flow mediated dilation procedure
Peak systolic tissue velocity | 12 months
  systolic tissue Doppler velocity assessed during resting and stress echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, prof, Study Director — Norwegian University of Science and Technology
Locations (2):
- University of Queensland, Brisbane, Australia
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Background] Dias KA, Coombes JS, Green DJ, Gomersall SR, Keating SE, Tjonna AE, Hollekim-Strand SM, Hosseini MS, Ro TB, Haram M, Huuse EM, Davies PS, Cain PA, Leong GM, Ingul CB. Effects of exercise intensity and nutrition advice on myocardial function in obese children and adolescents: a multicentre randomised controlled trial study protocol. BMJ Open. 2016 Apr 4;6(4):e010929. doi: 10.1136/bmjopen-2015-010929. PMID 27044585
- [Result] Dias KA, Ingul CB, Tjonna AE, Keating SE, Gomersall SR, Follestad T, Hosseini MS, Hollekim-Strand SM, Ro TB, Haram M, Huuse EM, Davies PSW, Cain PA, Leong GM, Coombes JS. Effect of High-Intensity Interval Training on Fitness, Fat Mass and Cardiometabolic Biomarkers in Children with Obesity: A Randomised Controlled Trial. Sports Med. 2018 Mar;48(3):733-746. doi: 10.1007/s40279-017-0777-0. PMID 28853029
- [Result] Ingul CB, Dias KA, Tjonna AE, Follestad T, Hosseini MS, Timilsina AS, Hollekim-Strand SM, Ro TB, Davies PSW, Cain PA, Leong GM, Coombes JS. Effect of High Intensity Interval Training on Cardiac Function in Children with Obesity: A Randomised Controlled Trial. Prog Cardiovasc Dis. 2018 Jul-Aug;61(2):214-221. doi: 10.1016/j.pcad.2018.01.012. Epub 2018 Feb 13. PMID 29452134
- [Derived] Dias KA, Ramos JS, Wallen MP, Davies PSW, Cain PA, Leong GM, Ingul CB, Coombes JS, Keating SE. Accuracy of Longitudinal Assessment of Visceral Adipose Tissue by Dual-Energy X-Ray Absorptiometry in Children with Obesity. J Obes. 2019 Nov 3;2019:2193723. doi: 10.1155/2019/2193723. eCollection 2019. PMID 31781386
- [Derived] Dias KA, Spence AL, Sarma S, Oxborough D, Timilsina AS, Davies PSW, Cain PA, Leong GM, Ingul CB, Coombes JS. Left ventricular morphology and function in adolescents: Relations to fitness and fatness. Int J Cardiol. 2017 Aug 1;240:313-319. doi: 10.1016/j.ijcard.2017.03.047. Epub 2017 Mar 11. PMID 28372865